CLINICAL TRIAL: NCT06474624
Title: Evaluation of the Effects of High-Intensity-Intermittent Training and Moderate-Intensity Continuous Training on Heart Rate Recovery, Functional Capacity, Fatigue and Quality of Life in Coronary Artery Patients
Brief Title: Evaluation of the Effects of Training at Different Intensities in Coronary Artery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Fatima Yaman, Principal Investigator, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-08/01
Record Dates: First submitted 2024-06-20; First posted 2024-06-25 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Coronary Heart Disease; Quality of Life; Functional Capacity; Fatigue
MeSH Terms: conditions — Coronary Disease; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity Continuous Training (Experimental): * A total of 24 -30 (8-10 weeks) sessions of an exercise-based Cardio Rehabilitation program 3 days a week.
  * Cycling for 20-30 minutes at 50-70% of Wmax between warm-up and cool-down periods.
  Interventions: Other: Cardio Rehabilitation program; Other: Cycling for 20-30 minutes
- High-intensity interval training (Experimental): * A total of 24 -30 (8-10 weeks) sessions of an exercise-based Cardiac Rehabilitation program 3 days a week.
  * Cycling a total of 4 cycles consisting of 4 minutes at 85-100% of Wmax followed by 3 minutes of active recovery periods at 50-70% of Wmax between warm-up and cool-down periods.
  Interventions: Other: Cardio Rehabilitation program; Other: Cycling a total of 4 cycles

INTERVENTIONS:
Other: Cardio Rehabilitation program — A total of 24 30 (8-10 weeks) sessions of an exercise-based Cardio Rehabilitation program 3 days a week.
Other: Cycling for 20-30 minutes — Cycling for 20-30 minutes at 50-70% of Wmax between warm-up and cool-down periods.
  Arms: Moderate Intensity Continuous Training
Other: Cycling a total of 4 cycles — Cycling a total of 4 cycles consisting of 4 minutes at 85-100% of Wmax followed by 3 minutes of active recovery periods at 50-70% of Wmax between warm-up and cool-down periods.
  Arms: High-intensity interval training

SUMMARY:
Coronary heart disease (CHD) remains the leading cause of morbidity and mortality in developed countries, accounting for approximately one-third of all deaths in individuals over 35 years of age.

Despite research to date, the basis of the disease is still poorly understood, with chronic dysfunction of the autonomic nervous system being proposed as such a basis, as well as pathophysiological and pathogenic approaches. Hypertension has been implicated in the development of cardiovascular risk factors such as diabetes and dyslipidaemia and is directly linked to mortality caused by coronary artery disease.

Moderate Intensity Continuous Training (MICT) has been recognised as the gold standard for many years. However, for some time, different researchers have adopted the high-intensity interval training model (HIIT) as the most effective method in terms of objective adaptations of most cardiac rehabilitation programmes in patients with coronary artery disease (CAD) and congestive heart failure.

High-intensity interval training (HIIT) consists of cycles between warm-up and cool-down periods, high-intensity exercise intensity followed by an active recovery period. The duration and intensity of these cycles vary between studies and there is no consensus on which is the optimal cycle. In general, the high-intensity exercise phase is applied at 80-100% of VO2 max and the active recovery phase is used between 50-70% of VO2 max.

In Moderate Intensity Continuous Training the submaximal exercise intensity determined in accordance with the patient's functional capacity between the warm-up and cool-down periods is applied for a fixed period. The Moderate Intensity Continuous Training is planned to consist of 20-30 minute sessions between 50-70% of maximum oxygen consumption (VO2max).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 30 and 65,
* Being with stable New York Heart Association functional class I or II coronary artery disease with angina pectoris or myocardial infarction,
* Having a left ventricular ejection fraction of 40% or above,
* Being clinically stable for more than 2 weeks in terms of symptoms and medical treatment.

Exclusion Criteria:

* Symptoms of ischaemia,
* Being in Class III-IV according to the New York Heart Classification,
* Presence of significant left ventricular outflow obstruction,
* Ventricular arrhythmia,
* Significant valvular heart disease,
* Failure to comply with the rules of exercise testing and training,
* Significant orthopaedic or neurological comorbidity preventing full participation.
* Less than 80% participation in the treatment programme
* Metabolic, haematological or other inflammatory diseases
* Known psychiatric illness
* Active malignancy and/or those diagnosed with malignancy within the last 5 years
* Those who have used tobacco products in the last 5 years
* BMI >35
* History of major orthopaedic surgery within the last 6 months.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Test (CPET) - Heart Rate Recovery | 8 weeks
  Cardiopulmonary exercise testing (CPET) is performed on patients with a bicycle ergometer, including analysis of exhaled gases. The testing protocol is tailored to the physical condition of each patient in gradual increments of 10, 15 or 20 W/min. The same protocol is used before and after the exercise training programme. The aim of exercise testing is to obtain a sustained effort for 8 to 12 minutes in order to maintain favourable oxygen uptake (VO2) kinetics and a linear relationship between VO2, exercise workload and heart rate (HR). A 12-lead ECG is continuously monitored and blood pressure is measured every 3 min during exercise tests. Resting heart rate, maximum heart rate, maximum load (watts), systolic blood pressure, diastolic blood pressure, VO2 max and/or VO2 estimate, HRR-1 and HRR-2 values are recorded before and after treatment as CPET data. HRR indices are calculated by subtracting the first and second-minute HR during the recovery period from the maximal HR.
Cardiopulmonary Exercise Test (CPET) - Functional Capacity | 8 weeks
  Cardiopulmonary exercise testing (CPET) is performed on patients with a bicycle ergometer, including analysis of exhaled gases. The testing protocol is tailored to the physical condition of each patient in gradual increments of 10, 15 or 20 W/min. The same protocol is used before and after the exercise training programme. The aim of exercise testing is to obtain a sustained effort for 8 to 12 minutes in order to maintain favourable oxygen uptake (VO2) kinetics and a linear relationship between VO2, exercise workload and heart rate (HR). A 12-lead ECG is continuously monitored and blood pressure is measured every 3 min during exercise tests. Resting heart rate, maximum heart rate, maximum load (watts), systolic blood pressure, diastolic blood pressure, VO2 max and/or VO2 estimate, HRR-1 and HRR-2 values are recorded before and after treatment as CPET data. HRR indices are calculated by subtracting the first and second-minute HR during the recovery period from the maximal HR.

SECONDARY OUTCOMES:
Fatigue Severity Scale | 10 weeks
  In the scale consisting of nine items that patients can self-administer, each item is scored between 1-7 (1=strongly disagree, 7=strongly agree) and questions the fatigue status in the last month. The scale score is the average value of the questions. If the average score is 5 and above, it is considered as "there is fatigue". An increase in the scale score indicates an increase in the level of fatigue.
36-Item Short Form Survey (SF-36) | 10 weeks
  It was developed by Ware et al. in 1992. The survey consists of a total of 36 questions with sub-headings such as function, role limitations related to physical health, role limitations related to emotional health, social function, mental health, energy, body pain, perception of general health and health change. The person can evaluate both negative and positive aspects of the health status. The total score varies between 0 and 100. A lower total score indicates a worse health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya University of Health Sciences Evliya Çelebi Physical Medicine and Rehabilitation Clinic, Cardiopulmonary Rehabilitation Unit, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No